CLINICAL TRIAL: NCT01033578
Title: Efficacy of Postoperative Adjuvant Treatments After Hepatectomy and Thrombectomy for Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis
Brief Title: Efficacy of Postoperative Adjuvant Treatments for Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Jia Fan, Liver Cancer Institute, Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fudan-LCI-PVTT-1
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): Receive hepatectomy and thrombectomy alone, no postoperative adjuvant treatments
  Interventions: Other: PVIC, TACE
- PVIC Group (Experimental): Portal Vein Infusion Chemotherapy (PVIC): 5-fluorouracil (650 mg/m2 for 24 hours on days 1), doxorubicin (10 mg/m2 for 6 hours on days 2), and cisplatin (20 mg/m2 for 6 hours on days 3) was continuously infused into portal vein through tube by a infusion pump implanted in operation. Treatment started 2 weeks after the operation and was repeated every 4 weeks for six cycles.
  Interventions: Other: PVIC, TACE
- TACE Group (Experimental): Transcatheter Arterial Chemoembolization (TACE): 5-fluorouracil (650 mg/m2), doxorubicin (10 mg/m2), cisplatin (20 mg/m2), and lipiodol 5ml were injected into hepatic artery by puncturing the common femoral artery in the right groin and passing a catheter through the abdominal aorta, through the celiac axis and common hepatic artery, into the proper hepatic artery. Treatment started 4 weeks after the operation and was repeated at 6-8 weeks intervals for 3 cycles.
  Interventions: Other: PVIC, TACE
- PVIC+TACE Group (Experimental): Combination of PVIC and TACE. PVIC started 2 weeks after operation and TACE started 6 weeks after operation. Both PVIC and TACE were repeated at 8 weeks intervals for 3 cycles.
  Interventions: Other: PVIC, TACE

INTERVENTIONS:
Other: PVIC, TACE — PVIC：5-fluorouracil (650 mg/m2 for 24 hours on days 1), doxorubicin (10 mg/m2 for 6 hours on days 2), and cisplatin (20 mg/m2 for 6 hours on days 3) were continuously infused into portal vein through tube by a infusion pump. Treatment started 2 weeks after the operation and was repeated every 4 weeks for 6 cycles.
  TACE: 5-fluorouracil (650 mg/m2), doxorubicin (10 mg/m2), cisplatin (20 mg/m2), and lipiodol 5ml were injected into hepatic artery by puncturing the common femoral artery in the right groin and passing a catheter through the abdominal aorta, through the celiac axis and common hepatic artery, into the proper hepatic artery. Treatment started 4 weeks after the operation and was repeated at 6-8 weeks intervals for 3 cycles.
  Other Names: PVIC: portal vein infusion chemotherapy; TACE: transcatheter arterial chemoembolization

SUMMARY:
The aim of this study is to assess efficacy of the different adjuvant chemotherapy strategies after hepatectomy and thrombectomy for hepatocellular carcinoma (HCC) and portal vein tumor thrombosis( PVTT).

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the sixth most common cancer worldwide and the third major cause of cancer-related death. HCC is characterized by its propensity for portal vein invasion. Portal vein tumor thrombosis (PVTT) can be detected macroscopically in the portal vein in 44% to 62.2% of autopsy cases. The natural history of untreated HCC with PVTT is dismal. The median survival of such patients was reported to be 2.7 mouths.

Non-surgical therapies, such as systemic/regional chemotherapy and transcatheter arterial embolization / transcatheter arterial chemoembolization (TAE/TACE), are not effective in treating HCC with PVTT. With the improvement of surgical techniques, surgical resection has been reported to achieve promising results. However, the high rate of recurrence and metastasis constitutes one of the most important challenges in improving surgical efficacy for HCC with PVTT.

There is rare report about prevention and treatment of postoperative recurrence and metastasis for HCC with macroscopical PVTT patients. We previously found the postoperative portal vein infusion chemotherapy (PVIC) and TACE benefited PVTT patients, which required further prospective randomized controlled studies with large case number to support our findings. The randomized controlled trial was design to investigate the efficacy of the different adjuvant chemotherapy strategies after hepatectomy and thrombectomy for HCC and PVTT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years
2. Hepatocellular carcinoma with portal vein tumor thrombosis in the first branch and/or main trunk of the portal vein confirmed by preoperative radiologic investigations, intraoperative exploration and postoperative pathology.
3. No extrahepatic metastasis
4. No previous management
5. The tumor and PVTT were completely removed confirmed by macroscopy and intraoperative ultrasonography
6. Good or moderate hepatic function (Child-Pugh Class A or B)
7. Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less

Exclusion Criteria:

1. Refuse to participate
2. Absolute neutrophil count <1.5*109/L, hemoglobin < 80g/L or platelet count <50 * 109/L, transaminases greater than 3 times the upper limit of normal, serum creatinine greater than 1.5 times the upper limit of normal, INR greater than 1.5 times of normal, which could not recover after treatment
3. Ascites refractory to diuretics
4. Variceal bleeding
5. Severe diseases of the heart or Lung

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 1999-10; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 1-year, 3-year, 5-year

SECONDARY OUTCOMES:
Time to Recurrence | 1-year, 3-year, 5-year

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, Doctor, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Liver Cancer Insitute, Zhongshan Hospital, Shanghai, China